CLINICAL TRIAL: NCT05202288
Title: Phase IIa, Randomized, Open-label, Parallel-group Trial to Assess the Immunogenicity, Safety and Tolerability of Ervebo Vaccine Administered With Inmazeb to Healthy Adult Volunteers.
Brief Title: Impact of Delay Between Administration of Inmazeb Administration and Vaccination by Ervebo on Vaccine Immune Response on Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: University of Bordeaux (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Clinical and Operational Research Alliance (CORAL) (Unknown); Institut Pasteur (Industry); Regeneron Pharmaceuticals (Industry); MSD France (Industry); Alliance for International Medical Action (Other); Centre de Recherche et de Formation en Infectiologie de Guinée (CERFIG) (Unknown); PACCI Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANRS 0064S IMOVA
Record Dates: First submitted 2021-12-15; First posted 2022-01-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Ebola Virus Disease
Keywords: Post Exposure Prophylaxis; Ebola vaccine
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — atoltivimab, maftivimab, and odesivimab-ebgn drug combination

STUDY DESIGN:
Intervention Model Description: The trial will have 6 arms:
  A control arm of vaccination alone will serve to characterize the immune response to the vaccine and it will be used as a comparator of vaccine immune response in the intervention arms. A control arm of mAb alone will serve to characterize the pharmacokinetic profile of mAb in the Guinean population. The 4 arms including different doses of Inmazeb plus vaccination were designed to mimic a time interval between Ervebo and Inmazeb administration (15, 57 and 169 days after Inmazeb).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Ervebo 72 million PFU (Active Comparator): The control arm (vaccination alone) will serve to characterize the immune response to the vaccine and it will be used as a comparator of vaccine immune response in the intervention arms. Administration at D1.
  Interventions: Biological: Ervebo
- Inmazeb 150mg/kg (Active Comparator): This second control arm of mAb alone will serve to characterize the pharmacokinetic profile of mAb in the Guinean population. Administration at D1.
  Interventions: Drug: Inmazeb
- Inmazeb 150mg/kg + Ervebo 72 million PFU (Experimental): The Arm 3, is a concomitant administration of the antibody and the vaccine at D1.
  Interventions: Biological: Ervebo; Drug: Inmazeb
- Inmazeb 50mg/kg + Ervebo 72 million PFU (Experimental): The Arm 4, is a concomitant injection of different-dose of the antibody and the vaccine. This design mimics a time interval of 15 days between Ervebo and Inmazeb administration. The administration will be at D1.
  These may help define a time interval between Ervebo administration and Inmazeb infusion.
  Interventions: Biological: Ervebo; Drug: Inmazeb
- Inmazeb 10mg/kg + Ervebo 72 million PFU (Experimental): The Arm 5, is a concomitant injection of different-dose of the antibody and the vaccine. This design mimics a time interval of 57 days between Ervebo and Inmazeb administration. The administration will be at D1.
  These may help define a time interval between Ervebo administration and Inmazeb infusion.
  Interventions: Biological: Ervebo; Drug: Inmazeb
- Inmazeb 0.7mg/kg + Ervebo 72 million PFU (Experimental): The Arm 6, is a concomitant injection of different-dose of the antibody and the vaccine. This design mimics a time interval of 169 days between Ervebo and Inmazeb administration. The administration will be at D1.
  These may help define a time interval between Ervebo administration and Inmazeb infusion.
  Interventions: Biological: Ervebo; Drug: Inmazeb

INTERVENTIONS:
Biological: Ervebo — Administration of r-VSV-ZEBOV vaccine
  Other Names: r-VSV-ZEBOV vaccine
  Arms: Ervebo 72 million PFU; Inmazeb 0.7mg/kg + Ervebo 72 million PFU; Inmazeb 10mg/kg + Ervebo 72 million PFU; Inmazeb 150mg/kg + Ervebo 72 million PFU; Inmazeb 50mg/kg + Ervebo 72 million PFU
Drug: Inmazeb — Administration of Inmazeb
  Other Names: REGN-E3B
  Arms: Inmazeb 0.7mg/kg + Ervebo 72 million PFU; Inmazeb 10mg/kg + Ervebo 72 million PFU; Inmazeb 150mg/kg; Inmazeb 150mg/kg + Ervebo 72 million PFU; Inmazeb 50mg/kg + Ervebo 72 million PFU

SUMMARY:
Ebola virus disease (EVD) is emerging regularly in various African countries for various reasons: during contact with mortal remains, during an unsafe burial or following the viral dissemination around a recovered patient.

However, tools to fight the spread of the disease are being made available to countries affected by EVD. A vaccine (Ervebo), developed by the Merck laboratory, demonstrated its efficacy in protecting contacts and contacts of contacts in the "Ebola That's Enough" trial and two monoclonal antibodies (Mabs) have demonstrated their efficacy in reducing mortality in patients with EVD: REGN-E3B (Inmazeb) and Mab114 (Ebanga).

The question of their use in post-exposure prophylaxis (PEP), defined as the treatment of contacts at very high risk of contracting EVD, is essential. Vaccination with Ervebo does not appear to be a good standalone option for PEP, particularly because antibody synthesis is delayed, and the vaccine is likely to be inactive for 10 days after administration. Monoclonal antibodies, on the other hand, seem to be a promising avenue in this indication because of their rapid action on the inhibition of virus entry into the cell.

Moreover, Ervebo vaccine expresses the viral target recognized by mAbs, GP EBOV. It is therefore possible that the vaccine response (production of vaccine antibodies) is inhibited by mAbs, which bind to GP EBOV and prevent vaccine replication, particularly in the case of concomitant administration.

However, no data on vaccine efficacy in combination are available. The question of the interaction between the monoclonal antibody and Ervebo and the delay between the administration of these two strategies remains unresolved.

The hypothesis of this trial is that Ervebo vaccine efficacy is diminished with the concomitant administration of a monoclonal antibody, especially if this administration is close (short time between Mabs and vaccination). We hypothesize that with an optimal delay between Mabs and vaccination, the immunogenicity of the vaccine when administered with monoclonal antibodies could be non-inferior to the vaccine alone, thus providing optimal short and long term protection.

The main objective of this study is to evaluate the extent of effect, if any, of Inmazeb administration on vaccine-induced neutralizing antibody responses to Zaire Ebola virus by Ervebo vaccine. If an interaction is observed, this will possibly enable determination of the time interval required between the administration of Inmazeb and Ervebo vaccine.

The trial will have 6 arms. A control arm of vaccination alone will serve to characterize the immune response to the vaccine and it will be used as a comparator of vaccine immune response in the intervention arms. A control arm of mAb alone will serve to characterize the pharmacokinetic profile of mAb in the Guinean population. The 4 arms including different doses of Inmazeb plus vaccination were designed to mimic a time interval between Ervebo and Inmazeb administration (15, 57 and 169 days after Inmazeb).

DETAILED DESCRIPTION:
Ebola virus disease (EVD) is emerging regularly in various African countries for various reasons: during contact with mortal remains, during an unsafe burial or following the viral dissemination around a recovered patient. In Guinea, 5 years after the end of the 2014-2016 epidemic that killed 11,000 people, a new epidemic has been declared in the southeast of the country and in Conakry in early 2021. In the Democratic Republic of Congo (DRC), the thirteenth epidemic was declared in early October 2021 in North Kivu province. However, more and more tools to fight the spread of the disease are being made available to countries affected by EVD. During the 2014 West African epidemic, a vaccine (Ervebo), developed by the Merck laboratory, demonstrated its efficacy in protecting contacts and contacts of contacts in the "Ebola That's Enough" trial. This vaccine has since been widely used as part of ring vaccination strategies during the most recent epidemics (2018-2021) in the DRC and the epidemic in Forest Guinea in 2021. In addition, during the tenth DRC epidemic (2018-2020), a compassionate trial (MEURI) and then a randomized controlled therapeutic trial was evaluating 4 molecules (3 passive immunotherapies and 1 direct antiviral) as a specific treatment for EVD. Two monoclonal antibodies (Mabs) have demonstrated their efficacy in reducing mortality in patients with EVD: REGN-E3B and Mab114.

With the availability of these management and prevention tools, the question of their use in post-exposure prophylaxis (PEP), defined as the treatment of contacts at very high risk of contracting EVD, is more essential than ever. Indeed, it seems clear that PEP is one of the major axes to be deployed to effectively control EVD. Several PEP strategies have therefore been discussed. Vaccination with Ervebo does not appear to be a good standalone option for PEP, particularly because antibody synthesis is delayed, and the vaccine is likely to be inactive for 10 days after administration. On the other hand, monoclonal antobodies seem to be a promising in this indication because of their rapid action on the inhibition of virus entry into the cell or on the virus itself, both in animal models and in humans.

However, while monoclonal antibodies are good candidates for PEP, they certainly do not provide sustained immunity. Specifically, in high-risk contacts with EVD, PEP with use of mAbs may allow them to avoid the infection associated with that specific contact, but not the persistent risk of infection during the epidemic. Therefore, vaccination is also necessary.

Moreover, Ervebo vaccine expresses the viral target recognized by mAbs, GP EBOV. It is therefore possible that the vaccine response (production of vaccine antibodies) is inhibited by mAbs, which bind to GP EBOV and prevent vaccine replication, particularly in the case of concomitant administration. However, no data on vaccine efficacy in combination are available. The question of the interaction between the monoclonal antibody and Ervebo and the delay between the administration of these two strategies remains unresolved.

The hypothesis of this trial is that vaccine efficacy is diminished with concomitant administration of a monoclonal antibody, especially if this administration is close (short time between Mabs and vaccination). We hypothesize that with an optimal delay between Mabs and vaccination, the immunogenicity of the vaccine combined with monoclonal antibodies could be non-inferior to that of the vaccine alone, thus providing optimal short and long term protection.

The trial will have 6 arms. A control arm of vaccination alone will serve to characterize the immune response to the vaccine and it will be used as a comparator of vaccine immune response in the intervention arms. A control arm of mAb alone will serve to characterize the pharmacokinetic profile of mAb in the Guinean population. The 4 arms including different doses of Inmazeb plus vaccination were designed to mimic a time interval between Ervebo and Inmazeb administration (15, 57 and 169 days after Inmazeb).

From an operational point of view, the ideal solution would be to be able to administer the vaccine at the same time as the Mab (simultaneous arm) or as soon as possible after the Mab is administered. Indeed, when implementing a PEP strategy during an epidemic, delaying vaccination represents a double risk for the patient: i) not being protected between the end of the Mab action and the vaccine and ii) not receiving the vaccine at all due to lack of compliance because of the long delay between contact and vaccination. The early, intermediate and late arms of the IMOVA trial will therefore assess the immunological response when the vaccine is administered 15, 57 or 169 days after Mab and thus determine the optimal time between the two interventions. For this purpose, the vaccine response will be analyzed in order to be put in perspective with the acceptable operational delay to guarantee protection and patient compliance.

The trial will take place in Guinea, in Conakry during a non-epidemic period for EVD on healthy volunteers. Indeed, it is important that participants in the IMOVA trial are not exposed to Ebola virus during their follow-up, to ensure the absence of potential infection in the late arms in particular. Therefore, if an epidemic were to occur in Guinea, enrollment in the IMOVA trial would be immediately halted and be restarted at the end of the epidemic period. The National Health Research Ethics Committee of Guinea (CNERS) will of course be informed of such a situation

ELIGIBILITY:
Inclusion Criteria:

* Available for the duration of the protocol follow-up;
* Consent to participate ;
* Agreed not to participate in another clinical research study until the end of the trial follow-up.

Exclusion Criteria:

* Prior history of EVD (self-reported);
* Previous vaccination with r-VSV-ZEBOV or any other Ebola vaccine (self-reported);
* Previous administration of Ebola antibody;
* HIV-1 and/or 2 positive serology;
* Pregnant women (positive pregnancy test);
* Breastfeeding women;
* To the opinion of the investigator, any clinically significant acute/chronic condition that would limit the participant's ability to meet the requirements of the study protocol;
* Taking Immunosuppressive therapy;
* Participation in another clinical research study within the last 30 days;
* Allergy to any component of the vaccine or Mabs;
* Person deprived of freedom by a judicial or administrative decision;
* Any other reason that, at the investigator's discretion, would compromise the participant's safety and cooperation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Neutralizing antibodies rates | Day 1, Day 29, Day 57, Day 85 and during participant's early termination
  The level will be evaluated with a pseudo-type plaque reduction neutralization test

SECONDARY OUTCOMES:
Anti-EBOV GP IgG rates | Day 1, Day 29, Day 57, Day 85 and during participant's early termination
  Measurement of EBOV GP IgG rate with the FANG technique
RT-PCR VSV | Day 3
  Standard biology
T cell response | Day 1, Day 29
  Performed by Intracellular Cytokine Staining (ICS)
Proportion of participants with grade 3 or 4 adverse events | Day 3, Day 7, Day 29, Day57, Day 85 and anytime after infusion and vaccination
  Proportion of participants with grade 3 or 4 adverse events
Proportion of participants lost to follow-up | Day 85 after vaccination
  Proportion of participants lost to follow-up
PK assessments | Day 1,Day 3, Day 29, Day 57, Day 85 and during participant's early termination
  Pharmacokinetics will be assessed by measuring the PK variable is the concentrations of REGN3470, REGN3471 and REGN3479 in serum over time.
Anti-Drug Antibodies (ADA) | Day 1, Day 85 and during participant's early termination
  measure of the immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Marie JASPARD, PHD, Principal Investigator — CORAL

IPD SHARING:
Plan to Share IPD: No